CLINICAL TRIAL: NCT05626218
Title: Effect of Stress Ball Application on Anxiety Pregnancy During the Non-stress Test: Experimental Study With Randomized Control
Brief Title: Application of Stress Ball and Non-stress Test With Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssistant professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliAS-7
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anxiety; Pregnancy Related
Keywords: anxiety; pregnancy; stress ball; non-stress test
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball group (Experimental): A stress ball will be applied to pregnant women with anxiety during NST.
  Interventions: Other: stress ball
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce anxiety symptoms.

INTERVENTIONS:
Other: stress ball — The woman is usually laid in the last side position during the procedure. A stress ball will be given to the right hand of the participants during the NST procedure (average 15-20 minutes). This stress ball will be squeezed for 2-3 seconds, and then the hand and arm will be told to relax. This process will be repeated throughout the NST. Hospital protocol will also be applied to these participants.
  Arms: Stress ball group

SUMMARY:
This research was planned as a randomized controlled experimental study to reduce the anxiety expectant mothers feel when on a non-stress test.

DETAILED DESCRIPTION:
Fetal well-being is assessed by evaluating fetal heart rate (FHR) patterns. The primary aim is to identify fetuses at risk of intrauterine death or neonatal complications and, if possible, intervene (usually by delivery) to prevent these adverse outcomes. The most commonly used method for this purpose is the non-stress test. Non-stress test (NST) is a non-invasive fetal evaluation method. The NST is evaluated for at least 20 minutes while the expectant mother is lying supine or left-side.

Although it is a painless procedure, it takes about 20 minutes, and the pregnant woman stays in the same position throughout the procedure, creating although there are many methods to reduce stress, it is thought that a cheap and easily accessible stress ball can be used as a method of distraction or distraction. Although there are studies investigating the effectiveness of stress balls in managing various disease groups and symptoms in the literature, no study has been found to examine the NST effectiveness of stress balls. This research was planned as a randomized controlled experimental study to reduce the stress felt by women who had a non-stress test during pregnancy by applying a stress ball during the procedure. anxiety for the pregnant woman. The fact that the pregnant woman has high anxiety during the procedure affects the test result and may increase the false-positive rate and cause false evaluation. This increase in the false-positive rate in NST results may lead to an increase in an operative delivery. However, it is the midwives' responsibility to eliminate the situations that cause anxiety in pregnant women, which may affect the NST result before and during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand Turkish
* Being between the ages of 20-35
* Single pregnancy
* Having had NST before

  ¬- Have eaten at least 2 hours before the NST procedure
* Don't be primiparous
* Getting 37 or less on the trait anxiety (STAI-1) scale
* Getting 37 or more on the state anxiety (STAI-2) scale
* Volunteering to participate in the research
* Fully answering survey and scale forms
* Being in the 3rd trimester

Exclusion Criteria:

* Having been diagnosed with a risky pregnancy
* Unwilling to continue working
* Having a chronic disease (Diabetes, Hypertension, Thyroid etc.),
* Having any problem that prevents communication (such as hearing, speaking, and understanding abilities),
* Using one of the pharmacological or non-pharmacological methods to reduce stress and receiving psychiatric treatment (Pharmacotherapy or psychotherapy).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Introductory Information form | between one to six months
  A form that includes questions about women's socio-demographic and pregnancy and characteristics.
  A form that includes questions about women's socio-demographic and pregnancy and characteristics.
the Spielberger State-Trait Anxiety Inventory (STAI/1-2) scale | between one to six months
  This scale, developed by Spielberg in 1973, consists of 40 questions. It is a 4-point Likert type scale (1=not at all, 4=very much). The lowest score that can be obtained from the scale is 20, and the highest score is 80. The higher the score is, the higher the anxiety level is. The alpha value of the scale is 0.86-.92.33. The validity and reliability study in our country was conducted by Oner et al., in 1983 and the alpha value was found between. The scale that will be used to evaluate the state and trait anxiety of pregnant women. As the score increases, it is determined that the anxiety is higher.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Dağlı, Phd, Principal Investigator — Cukurova University; AYCA SOLT KIRCA, Phd, Study Director — Kırklareli University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)